CLINICAL TRIAL: NCT01948804
Title: The Comparison of Effect of Four Different Treatment Protocols: Antagonist/Letrozole Protocol, Microdose Flare-up Protocol, Antagonist/Clomiphene Protocol, Antagonist on IVF Outcomes in Poor Responders Undergoing in Vitro Fertilization; a Prospective Randomized-controlled Study.
Brief Title: The Comparison of Effect of Four Different Treatment Protocols on IVF Outcomes in Poor Responders Undergoing in Vitro Fertilization.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Pınar Özcan Cenksoy (Other)
Responsible Party: Sponsor-Investigator, Pınar Özcan Cenksoy, Medical Doctor, Yeditepe University Hospital
Organization: Yeditepe University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ytu-123; ytu-123 (Other: YeditepeUH)
Record Dates: First submitted 2013-09-06; First posted 2013-09-24 (Estimated); Last update posted 2014-01-15 (Estimated); Status verified 2014-01

CONDITIONS: Poor Responders Undergoing IVF
MeSH Terms: interventions — cetrorelix; Letrozole; Leuprolide; follitropin alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IVF patients (Experimental): patients that has applied to Yeditepe University Hospital assisted reproduction center
  Interventions: Drug: GnrH Antagonist/letrozole protocol (Cetrotide; serono + Femara; Novartis Pharma AG); Drug: microdose flare-up protocol (Lucrin; Abbott + Gonal F, Serono); Drug: Antagonist/clomiphene protocol (Cetrotide; serono + Klomen, Kocak pharma); Drug: GnRH antagonist protocol (Cetrotide, Serono)

INTERVENTIONS:
Drug: GnrH Antagonist/letrozole protocol (Cetrotide; serono + Femara; Novartis Pharma AG)
Drug: microdose flare-up protocol (Lucrin; Abbott + Gonal F, Serono)
Drug: Antagonist/clomiphene protocol (Cetrotide; serono + Klomen, Kocak pharma)
Drug: GnRH antagonist protocol (Cetrotide, Serono)

SUMMARY:
The comparison of effect of four different treatment protocols: Antagonist/letrozole protocol, microdose flare-up protocol, Antagonist/clomiphene protocol, Antagonist on IVF outcomes in poor responders undergoing in vitro fertilization; a prospective randomized-controlled study.

ELIGIBILITY:
Inclusion Criteria:

Criteria for definition of poor responders included at least one of the following

1. Anti müllerian hormone <1.1 ng/ml and/or a previous poor ovarian response (≤3 oocytes with a conventional stimulation protocol).
2. Primary infertile patients
3. BMI≤30 kg/m2 were included this study.

Exclusion Criteria:

-

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-01; Primary Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
clinical pregnancy rates | 6 months

SECONDARY OUTCOMES:
total number of oocytes retrieved | 6 months